CLINICAL TRIAL: NCT04876131
Title: CHOICE UTI - Clinical Efficacy of Single Dose (Daily) IV Antibiotics Followed by 2 Days Oral Antibiotics Compared to 3 Doses (Daily) IV Antibiotics for Children With Complicated Urinary Tract Infections: a Multicentre Randomised Trial
Brief Title: Single Dose Intravenous Antibiotics for Complicated Urinary Tract Infections in Children
Acronym: CHOICE UTI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72065
Record Dates: First submitted 2021-05-02; First posted 2021-05-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: Complicated Urinary Tract Infection; Infection; Pediatric Infectious Disease
MeSH Terms: conditions — Infections | interventions — Penicillin G; Gentamicins; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Participants will be recruited when they present to the emergency department with a complicated UTI. Once they have been consented to the study they will then be randomised into one of the treatment arms, these treatment arms will run parallel to one another.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1, 1 dose (Experimental): * Single dose IV to cover Gram negative bacteria followed by 2 days of oral antibiotics
  * Single dose IV to cover Enterococcus spp
  IV antibiotics are as per local institutional guidelines and microbiology eg: IV gentamicin with or without IV benzylpenicillin. Gentamicin is used when Gram Negative coverage is appropriate, benzylpenicillin is also used when Enterococcus coverage is appropriate, depending on local microbiology data. Once the IV component is complete the patient will be given an oral antibiotic (cefalexin) on day 2 and 3 of the study.
  Interventions: Drug: Benzylpenicillin - single dose; Drug: Gentamicin - single dose; Drug: Cefalexin - post single dose of IV antibiotics for the remaining two days
- Arm 2, 3 doses (Active Comparator): * 3 doses IV to cover Gram negative bacteria
  * 3 days IV antibiotics to cover Enterococcus spp
  IV antibiotics are as per local institutional guidelines and microbiology eg: IV gentamicin with or without IV benzylpenicillin. Gentamicin is used when Gram Negative coverage is appropriate, benzylpenicillin is also used when Enterococcus coverage is appropriate, depending on local microbiology data.
  Interventions: Drug: Benzylpenicillin - three days; Drug: Gentamicin - three days

INTERVENTIONS:
Drug: Benzylpenicillin - single dose — Participants will receive a single dose of IV antibiotic (benzylpenicillin).
  Benzylpenicillin dosing: 1 month - 18 years, IV or Intramuscular (IM) 30 mg/kg (maximum 1.2 g) every 6 hours.
  Arms: Arm 1, 1 dose
Drug: Benzylpenicillin - three days — Participants will receive three days of this IV antibiotic (benzylpenicillin).
  Benzylpenicillin dosing: 1 month - 18 years, IV or Intramuscular (IM) 30 mg/kg (maximum 1.2 g) every 6 hours. For severe infections, use up to 60 mg/kg (maximum 2.4 g) every 4-6 hours.
  Arms: Arm 2, 3 doses
Drug: Gentamicin - single dose — Participants will receive a single dose of IV antibiotic (gentamicin).
  Gentamicin dosing: Children ≤10 years old: 7.5 mg/kg (maximum dose 320 mg) Children >10 years old: 6-7 mg/kg (maximum dose 560 mg)
  Arms: Arm 1, 1 dose
Drug: Gentamicin - three days — Participants will receive three days of this IV antibiotic (gentamicin).
  Gentamicin dosing: Children ≤10 years old: 7.5 mg/kg (maximum dose 320 mg) Children >10 years old: 6-7 mg/kg (maximum dose 560 mg)
  Arms: Arm 2, 3 doses
Drug: Cefalexin - post single dose of IV antibiotics for the remaining two days — Oral antibiotic will be as per local guidelines. i.e. Cefalexin 25mg/kg (maximum dosage 500mg) 4 times a day or 33mg/kg (maximum dosage 500mg) 3 times a day
  Arms: Arm 1, 1 dose

SUMMARY:
Urinary tract infections (UTI) are commonly encountered in children, with 7% diagnosed with at least one UTI by the age of 19 years. The evidence for treatment of uncomplicated UTI is clear; oral antibiotics are as good as intravenous (IV) antibiotics, usually for a total of 7 days. Complicated UTIs (cUTIs) on the other hand, are common reasons for hospital admissions for IV antibiotics and constitute a major burden for healthcare systems. There is considerable variation in care for children who present with UTI and have complicating features such as vomiting, dehydration, urological abnormalities or have a previous history of UTI. Australian and international guidelines lack clear, evidence-based recommendations to guide treatment in this group. Without gold standard evidence, these children will continue to receive unnecessary IV antibiotics, longer hospital stays and poorer health outcomes.

This multicentre, non-inferiority randomised trial will investigate if One dose - single dose of IV followed by 2 days oral antibiotics is as non-inferior to Three doses for children with UTI and co-existing complicating factors presenting to the Emergency Department (ED). In other words, this study will compare if a single dose of IV antibiotics plus two days oral antibiotics is as clinically effective as 3 doses antibiotics in resolving UTI symptoms at 72 hours after the first dose of IV antibiotics, for complicated UTIs in children presenting to the ED. All participants will receive a total of 7 days of antibiotics for the complicated urinary tract infection. If 1 dose IV and 2 days oral antibiotics is found to be as good as 3 days, the duration of IV antibiotics for complicated UTI can be reduced along with avoidance of the inherent risks of unnecessary hospital admission by administering a single IV dose in an outpatient/ED setting. On the other hand if a single IV dose results in prolonged symptoms or treatment failure, this will inform practice for the proportion of children who have a single dose of IV antibiotics in the ED and are sent home on oral antibiotics. Regardless of the outcome, this trial will inform clinical practice for complicated UTI to improve health outcomes for this group.

DETAILED DESCRIPTION:
Study design:

An open label, multi-centre, pragmatic, non-inferiority randomised controlled trial (RCT).

It will incorporate a two-arm, non-inferiority design with parallel groups and 1:1 allocation of children with ≥2 complicated features of UTI presenting to the ED in whom clinicians deem parenteral antibiotics are required.

Primary objective:

The primary objective of this trial is to compare whether 1 dose of a daily parenteral antibiotic followed by 2 days oral antibiotics is as clinically effective (non-inferior) in resolving UTI symptoms at 72 hours after the first IV dose, as 3 doses of a daily parenteral antibiotic for complicated urinary tract infections presenting to the ED.

Definition:

1 dose: one dose of a daily dose IV to cover Gram negative bacteria +/- one dose IV to cover Enterococcus spp. This will be followed by two days oral antibiotics.

3 doses: three doses of a daily dose IV to cover Gram negative bacteria +/- 3 days IV antibiotics to cover Enterococcus spp.

Secondary objectives:

The secondary objectives of this trial are to compare the following outcomes between the 1 dose and the 3 doses arms:

* Readmission due to persistent fever, vomiting, rigors, or clinical deterioration (e.g., poor feeding, dehydration) within 14 days of the initial dose of IV antibiotics.
* Readmission due to persistent fever, vomiting, rigors, or clinical deterioration (e.g., poor feeding, dehydration) within 1 month of the initial dose of IV antibiotics.
* Transfer from HITH/ambulatory care to ward care during admission within 72 hours of the initial dose of IV antibiotics.
* Time to resolution of fever/vomiting/rigors within 72 hours of the initial dose of IV antibiotics as reported by parents/guardian.
* Improvement as determined by parents/guardian at 72 hours after the first IV dose.
* Antiemetic use for 72 hours from the initial IV antibiotic dose.
* Duration of IV antibiotics (actually received by patient) from the first dose of IV antibiotics to last dose of IV antibiotics.
* Duration of oral antibiotics (actually received by patient) from the first dose of oral antibiotics (after IV antibiotics started) to last dose of IV antibiotics.
* Total duration of antibiotics: sum of duration of IV antibiotics and oral antibiotics.
* Recurrence of UTI within 14 days from the first dose of IV antibiotics.
* Recurrence of UTI within 1 month from the first dose of IV antibiotics.
* Complications of UTI from the initial IV antibiotics dose to 14 days after the initial dose.
* Adverse events from the initial IV antibiotics dose to 14 days after the initial dose.
* Quality of life (QoL) indicators on Day 1 of IV antibiotics (within 24 hours of initial IV antibiotics) and after Day 4 (72 hours up to Day 7).
* Parental QoL on Day 14.
* Cost-effectiveness - hospital administrative data on costs and patient/parents reported costs.
* Follow up microbiological urine culture after commencing IV antibiotics.
* Imaging reports - ultrasound or other imaging results will be collected for patients who have them performed.

Intervention:

Patients who are eligible for the study will be randomised to receive 1 dose of daily IV antibiotics followed by 2 days of oral antibiotics or 3 doses of daily IV antibiotics . All participants will receive a total of 7 days treatment with antibiotics for the complicated urinary tract infection.

Oral antibiotics will start as soon as able to tolerate, within 12 hours of the last IV dose for both arms.

Study methodology:

Enrolment and randomisation: During ED assessment, clinicians will identify patients with a suspected UTI and screen patients against eligibility criteria. The relevant clinical team at each site will receive standardized, study specific education based on centrally developed study education materials. Presence of the following symptoms/sign will be recorded at baseline (fever, vomiting, rigors, tachycardia). Participants will be randomised to one of the 2 arms after written informed consent is obtained.

Intervention Day 1:

The first dose of the antibiotics will be commenced in the ED. Care of the patient will be as per routine clinical care. Decision for admission to hospital and location of treatment (ambulatory/Hospital-in-the-Home care) will be determined by the treating clinician as per routine clinical care. Parents will be provided with a thermometer and a diary to record a daily assessment of their child (fever, rigors, vomiting).

Intervention Day 4 :

72 hours after the first dose of IV antibiotics, a research nurse/assistant will conduct an assessment over phone or telehealth to obtain the primary outcome data: Persistence of baseline symptoms (fever, vomiting, rigors) or development of these symptoms (if not previously present) since baseline. Any ambiguity with regards to symptoms being attributable to UTI will be judged by a blinded clinician external to the research team.

Follow up Day 14:

14 days after the first dose of IV antibiotics, a research nurse/assistant will conduct an assessment over phone or telehealth for follow up data including whether GP/ED visit or readmission occurred for UTI and total duration of antibiotics taken by the patient.

Follow up 1 month:

1 month after the first dose of IV antibiotics, a research nurse/assistant will conduct an assessment over phone or telehealth for follow up data including whether GP/ED visit or readmission occurred for UTI, total duration of antibiotics taken by the patient.

ELIGIBILITY:
Inclusion Criteria:

* 3 months (corrected age) to 18 years
* Fever (reported fever at home or measured fever of ≥38 degrees Celsius associated with the illness that triggered current ED presentation (eg fever may have been 18 hours prior to presentation but none since then because patient has been on maximal antipyretics - paracetamol or ibuprofen)
* Any of the following complicating features: Vomiting, Rigors, History of recurrent UTI, Urological abnormalities, Tachycardia
* Urine sample available (Urine culture must have been collected prior to or within an hour of antibiotic treatment, either at the GP or ED - in order to assess urine culture as per below).
* Abnormal urinary dipstick leucocyte esterase >1+ or nitrite positive OR ≥5 White Blood Cells (WBCs) per high-power field in centrifuged urine OR≥ 10 White Blood Cells (WBCs) per mm3 in uncentrifuged urine and bacteriuria with any bacteria per high-power field
* ED clinician determines the child requires treatment with IV antibiotics * In ED, only urine dipstick or urinalysis will be available. Once urine culture is available, to be included in the efficacy analysis, culture results must meet the following criteria: Positive urine culture result with no more than 2 species of microorganisms AND Spontaneously voided urine with ≥105 microorganisms per mL of urine or Suprapubic aspirate or urinary catheter with ≥104 microorganisms per mL of urine. In the absence of a positive urine culture, ultrasonographic findings supporting pyelonephritis (per reporting radiologist) will be accepted as evidence of a urinary tract infection.

Exclusion Criteria:

* Sepsis (requiring inotropic support or more than 20ml/kg of fluid bolus in Emergency Department)
* Known allergy to all once daily study drug options (gentamicin or ceftriaxone or amikacin)
* If the patient has another co-existing condition which requires (based on established evidence-based guidelines) more than 1 dose of IV antibiotics eg meningitis
* Known chronic renal failure or renal transplant patients
* Unrepaired posterior urethral valves
* Indwelling stent and fever
* Previously enrolled participants in the CHOICE UTI trial.
* No available oral antibiotic option for this UTI: urine culture result already available and multi-resistant organism with susceptibility only to IV antibiotics or known intolerance to oral antibiotics (previous UTI with multi-resistant organism not an exclusion)
* Previous IV antibiotics for same UTI episode eg interhospital transfer whereby significant time has passed since first dose IV
* Patients with clinically suspected renal abscess e.g., extreme renal tenderness, out of keeping with pyelonephritis (clinically determined).
* Clinician does not intend on prescribing a course of IV antibiotics but plans on only giving a single dose from the outset
* Recurrence of urinary tract infection within 2 weeks
* Unable to obtain consent
* Patient is pregnant

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 452 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2028-05-16 (Estimated); Study Completion 2028-05-16 (Estimated)

PRIMARY OUTCOMES:
Risk difference between 1 dose and 3 doses IV in the proportion of participants with clinical failure at 72 hours | 72 hours
  Clinical failure is defined as persistence of baseline symptoms (fever, vomiting or rigors) or development of new symptoms (fever, vomiting or rigors) attributable to UTI at 72 hours. Assessment of clinical failure to be conducted at least 6 hours after antipyretic. Presence of fever, vomiting, or rigors reported by parents within 6 hours of assessment will be recorded as present at assessment.

SECONDARY OUTCOMES:
Risk difference between 1 dose and 3 doses IV in the proportion of participants readmitted or attending the ED within 14 days of the initial dose of IV antibiotic. | 14 days
  Proportion of readmissions within 14 days of the initial dose of IV antibiotics due to persistent fever, vomiting, rigors, or clinical deterioration (eg poor feeding, dehydration) that can be attributable to the UTI
Risk difference between 1 dose and 3 doses IV in the proportion of participants readmitted or attending the ED within 1 month of the initial dose of IV antibiotics | 1 month
  Proportion of readmission within 1 month of the initial dose of IV antibiotics due to persistent fever, vomiting, rigors, or clinical deterioration (eg poor feeding, dehydration) that can be attributable to the UTI.
Risk difference between 1 dose and 3 doses IV in proportion of participants transferred from HITH or ambulatory care to ward care within 72 hours of initial dose of IV antibiotics. | 72 hours
  Proportions of participants transferred from HITH or ambulatory care to ward care within 72 hours of initial dose of IV antibiotics.
Risk difference between 1 dose and 3 doses IV in the proportion of participants with parental reported improvement | 72 hours
  Proportion of patients who are reported as 'generally improved/better' at 72 hours of the initial IV antibiotic dose. This will be reported via the daily diary completed by the parent on day 1, 2 and 3.
Mean difference between 1 dose and 3 doses IV in duration of IV antibiotics usage | 7 days
  Mean difference between 1 dose and 3 doses IV group in duration (number of days up to 1 decimal point) of IV antibiotics, i.e. mean time difference from first dose of IV antibiotics to last dose of IV antibiotics
Mean difference between 1 dose and 3 doses IV in duration of oral antibiotic usage. | 14 days
  Mean difference between 1 dose and 3 doses IV in the duration (number of days up to 1 decimal point) of oral antibiotics administered to patients, i.e mean time difference between last dose of IV antibiotics and the last dose of oral antibiotics.
Risk difference between 1 dose and 3 doses IV in the proportion of participants with recurrence of UTI symptoms within 14 days of initial dose of IV antibiotics | 14 days
  Risk difference between 1 dose and 3 doses IV in the proportion of participants with recurrence of UTI symptoms within 14 days of the first dose of IV antibiotics. Recurrence of symptoms depends on what symptoms the patient initially presented with but may be classified as recurrence of fever, vomiting, rigors or tachycardia.
Risk difference between 1 dose and 3 doses IV in the proportion of participants with recurrence of UTI symptoms within 1 month of initial dose of IV antibiotics | 1 month
  Risk difference between 1 dose and 3 doses IV in the proportion of participants with recurrence of UTI symptoms within 1 month of initial dose of IV antibiotics. Recurrence of symptoms depends on what symptoms the patient initially presented with but may be classified as recurrence of fever, vomiting, rigors or tachycardia.
Risk difference in the proportion of participants with complications within 14 days of initial dose of IV antibiotics | 14 days
  Risk difference in the proportion of participants with complications within 14 days of initial dose of IV antibiotics. Complications are defined as abscess, sepsis, meningitis from the initial IV antibiotics dose to 14 days after the initial dose that are attributable to the UTI as judged by a clinician.
Mean difference in the proportion of participants who experience at least one adverse event within 14 days of the initial dose of IV antibiotics | 14 days
  Mean difference in the proportion of participants who experience at least one adverse event within 14 days of the initial dose of IV antibiotics. An adverse event is described as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Risk difference between the 1 dose and 3 doses IV groups in the proportion of participants who experience an allergic reaction attributable to the antibiotics administered within 14 days of the initial dose of IV antibiotics | 14 days
  Risk difference in the proportion of participants who experience an allergic reaction attributable to the antibiotics administered within 14 days of the initial dose of IV antibiotics. An allergic reaction is classified as an overreactive immune system to a harmless substance known as an allergen in this case a medicinal (investigational) product.
Mean difference between 1 dose and 3 doses IV on the weighted total score of the Child Health Utility instrument administered within 24 hours after initial dose of IV antibiotics. | 24 hours
  The Child Health Utility instrument is a 9 item parent-rated, preference-weighted measure used to calculate quality adjusted life years for children. This survey consist of 9 questions asking how the child is feeling and questions about their activity levels. The minimum score is zero and the maximum score for this survey is 1 which indicates optimal health. This should be completed within 24 hours of initial IV antibiotics
Mean difference between 1 dose and 3 doses IV on the weighted total score of the Child Health Utility instrument administered between day 5-7 of initial dose of IV antibiotics | Day 5 to 7
  The Child Health Utility instrument is a 9 item parent-rated, preference-weighted measure used to calculate quality adjusted life years for children. This survey consist of 9 questions asking how the child is feeling and questions about their activity levels. The minimum score is zero and the maximum score for this survey is 1 which indicates optimal health. This should be completed between day 5 to 7 after initial IV antibiotics
Mean difference between 1 dose and 3 doses IV in the cost-effectiveness of treatment groups. | Day 14
  Mean difference between 1 dose and 3 doses IV in the cost-effectiveness of treatment. As judged by survey provided to the families asking about their out of pocket expenses or loss of productive work hours.
Risk difference between the 1 dose and 3 doses IV groups in the proportion of patients with bacterial growth in urine culture (day 0) | Day 0
  Risk difference between the 1 dose and 3 doses IV groups in the proportion of patients with bacterial growth: for example E.Coli, Enterococcus.
Risk difference between the 1 dose and 3 doses IV in the proportion of patients with bacterial growth in urine culture (Day 14) | Day 14
  Risk difference between the 1 dose and 3 doses IV groups in the proportion of patients with bacterial growth: for example E.Coli, Enterococcus.
Risk difference between the 1 dose and 3 doses IV group in the proportion of patients administered antiemetics | Up to day 3
  Risk difference between the 1 dose and 3 doses IV in the proportion of patients administered antiemetics (commonly used antiemetics in children are metoclopramide, domperidone, ondansetron and prochlorperazine). As determined by parent reported diary, completed daily for the first 3 days after enrolment.
Risk difference between the 1 dose and 3 doses IV group in the proportion of patients administered antipyretic or analgesia. | Up to day 3
  Risk difference between the 1 dose and 3 doses IV group in the proportion of patients administered antipyretic or analgesia (commonly used antipyretics and analgesia in children are paracetamol, ibuprofen, naproxen). As determined by parent reported diary, completed daily for the first 3 days after enrolment.
Risk difference between the 1 dose and 3 doses IV group in the proportion of patients with abnormal imaging. | Up to1 month
  Risk difference between the 1 dose and 3 doses IV group in the proportion of patients with Ultrasound reported abnormalities of the renal tract.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Ibrahim, Principal Investigator — Murdoch Childrens Research Institute; Penelope Bryant, Principal Investigator — Murdoch Childrens Research Institute
Locations (6):
- Australia (5):
  - Women and Children's Hospital, Adelaide, South Australia
  - University Hospital Geelong, Geelong, Victoria
  - Monash Health, Melbourne, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Washington
- Starship Children's Hospital, Auckland, Auckland Province, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this study will be available six months after publication of the results. The study protocol, analysis plan and consent forms will also be available. This will all be available by contacting Murdoch Children's Research Institute.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome
Access Criteria: Prior to this data being made available a data access agreement much be signed between the relevant parties and approval by the trial steering committee. Data will only be shared with recognised research institutions